CLINICAL TRIAL: NCT05254522
Title: Fever of Unknown Orgin Registry in Internal Medicine Unit and Infectious Disease Units
Acronym: FUO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.07.2018
Record Dates: First submitted 2022-02-09; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Fever of Unknown Origin
MeSH Terms: conditions — Fever of Unknown Origin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: not aplicable since it is a Registry — not aplicable since it is a registry

SUMMARY:
This registry has the aim to collect epidemiological and clinical data of classical FUO cases in Italian Internal medicine Dept. and in Italian Infection diseases Dept.

DETAILED DESCRIPTION:
In particular this registry intends to record clinical data observed, diagnostic methods used and the clinical evolution of classical FUO cases

ELIGIBILITY:
Inclusion Criteria:

* • fever (temperature > 38.3° C) found in several occasions of a duration exceeding 3, unable to make a diagnosis after a period of 3 days of hospitalization or after 3 out-patients visits in Internal Medicine Dept. or Infection Diseases Dept.

  * signed informed consent

Exclusion Criteria:

* • immunocompromised patients

  * patients in treatment with steroidi (prednisone > 0,5 mg/Kg/die per > 4 weeks), anti-TNF, ciclofosfamide, tacrolimus, everolimus, sirolimus, azatioprina, ciclosporina, micofenolato, metotrexate
  * neutropenic patients with less than 500 neutrofili/µL
  * HIV positive patients
  * nocosomial fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (in- or out-patients) with classical FUO hospitalised in Internal Medicine Dept. and in Infectious Diseases Dept.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To describe FUO cases collected | 6 moths
  To describe clinical evolution of classical FUO cases recording clinical data observed, diagnostic methods used.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA FONTANELLA, Study Director — FADOI FOUNDATION
Locations (1):
- ASUI di Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luzzati R, Zerbato V, Attard L, Virgili G, Cilli A, Zanier A, Libanore M, Segala D, Tedesco A, Bortolotti ME, Pontali E, Feasi M, Re A, Giarretta I, Pomero F, Zagarri E, Concia E, Dentali F, Manfellotto D, Campanini M; FADOI-FUO Study Group. Fever of unknown origin (FUO) FADOI-SIMIT Italian registry: can demographics, comorbidities, and clinical variables predict the etiology of classic FUO?-a prospective Italian study. Intern Emerg Med. 2025 Nov;20(8):2331-2340. doi: 10.1007/s11739-025-04084-1. Epub 2025 Aug 19. PMID 40828443